CLINICAL TRIAL: NCT05060692
Title: Changes of NLF in Serum of Long COVID Patients
Status: Completed | Type: Observational
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Laura de Boni, Dr., University Hospital, Bonn
Other Study IDs: 1
Record Dates: First submitted 2021-08-09; First posted 2021-09-29 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Clinical Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LONGCOVID: Patient with Long-COVID Syndrom
  Interventions: Diagnostic Test: Bloot testing
- CONTROLS: Healthy individials
  Interventions: Diagnostic Test: Bloot testing

INTERVENTIONS:
Diagnostic Test: Bloot testing — NFL measruments in serum

SUMMARY:
The study investigates the blood NFL levels in Long-COVID patients.

DETAILED DESCRIPTION:
The study investigates the blood NFL levels in Long-COVID patients.

ELIGIBILITY:
Long-COVID Syndrom

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Long-COVID-Syndrome
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Levels of NFL over a 1 year course of the Long-COVID Syndrom | 1 year
  see above

CONTACTS AND LOCATIONS:
Locations (1):
- Laura de Boni, Bonn, Germany

IPD SHARING:
Plan to Share IPD: No